CLINICAL TRIAL: NCT02428101
Title: Relation of Genetic Polymorphism of ABCG2 Gene And Occurrence of Oxaliplatin - Induced Peripheral Neuropathy in Patients With Gastrointestinal Tract Cancer
Brief Title: Oxaliplatin - Induced Peripheral Neuropathy in Patients With Gastrointestinal Tract Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Inas M Ahmed, PH, African Union,organization St. Abbsia, Cairo, Egypt, Ain Shams University
Other Study IDs: master(No.38)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Gastrointestinal Tract Cancer; Peripheral Neuropathy
MeSH Terms: conditions — Gastrointestinal Neoplasms; Peripheral Nervous System Diseases | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Genetic: polymorphism analysis

SUMMARY:
This study will examine DNA from Gastrointestinal Tract of cancer patients treated with oxaliplatin to look for a variation (mutation) of the ABCG2 gene that may lead to drug-induced peripheral neuropathy in certain patients.

The DNA will be extracted from patients' blood samples and are analyzed for the ABCG2 single nucleotide polymorphism (G34A - rs2231137 and A/A -rs3114018 genotypes) and correlated with peripheral neuropathy grades.

DETAILED DESCRIPTION:
Pharmacogenetic analysis/genotyping :

Genotyping is conducted via High Resolution Melting (HRM) TECHNIQUE, To confirm the genotyping results, the Polymerase chain reaction (PCR) product of the samples will be examine via direct sequencing using 3500 Genetic analyzer from ThermoFisher (applied biosystem) at two ABCG2 loci using the following PCR primers:

1-ABCG2 G34A - rs2231137

Forward :

5'-TGC AAT CTC ATT TAT CTG GAC TA-'3

Reverse :

5'-AAT GCC TTC AGG TCA TTG GA-'3

-Annealing temp :57 -Product size : 163

2- ABCG2 A/A - rs3114018

Forward :

5'- TGATGTTCCTTCAGCCACTG-'3

Reverse :

5'-TTGTGGAAACCTCACAAAAGTG-'3

- Annealing temp : 59 - Product size : 124

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal Tract Cancer patients treated with Oxaliplatin-containing chemotherapy
* Measurable disease
* Age of 18 years to 80 years

Exclusion Criteria:

* Pregnant women
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Oxaliplatin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Neurologic disease or patients with disease impairing the neurologic function affecting

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Gastrointestinal tract (GIT) Cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Correlation of single nucleotide polymorphisms of ABCG2 gene (G34A - rs2231137 and A/A -rs3114018 genotypes) with peripheral neuropathy grades, using the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE) | After 6 cycles of chemotherapy (each cycle is15 days), for six months
  Peripheral Neuropathy Toxicity will be assessed every cycle for six months using the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE). Patients will be assigned to 4 groups according to the grades of neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Inas M Moukhtar Ahmed, B.pharma, Principal Investigator — Faculty of Pharmacy, Ain Shams Universty; Lamia M El Wakeel, Assoc. Prof, Study Director — Clinical Pharmacy, Ain Shams University; Abdel Hady A Abdel Wahab, Professor, Study Chair — Biochemistry & Molecular biology,Cairo University; Amr S Saad, Assoc. Prof, Study Chair — Clinical Oncology, Ain Shams University; Raafat R Abdel-Malek, Assoc. Prof, Study Chair — clinical oncology, cairo university
Locations (1):
- Ain Shams University hospitals, Cairo, Abbasia, Egypt